## **Study Protocol**

# Low-dose decitabine for refractory prolonged isolated thrombocytopenia after hematopoietic cell transplantation

Vision 3.0

Aug. 07, 2017

ClinicalTrials.gov Identifier: NCT02487563

Principal Investigator

Yue Han, MD, PhD, hanyue@suda.edu.cn; Depei Wu, MD, PhD, wudepei@suda.edu.cn. Jiangsu Institute of Hematology, The First Affiliated Hospital of Soochow University, Suzhou 215006, China.

## **Table of Contents**

| Protocol amendments | 4 |
|-----------------------------------------------------------------|----|
| Protocol summary | 5 |
| Background | 7 |
| Refractory prolonged isolated thrombocytopenia after allogeneic | |
| hematopoietic cell transplantation | 7 |
| rhTPO for thrombocytopenia | 8 |
| Decitabine for thrombocytopenia after HCT | 8 |
| Reference | 10 |
| Rationale of this study | 12 |
| Study objectives | 12 |
| Primary objective and primary endpoint | 12 |
| Secondary objectives and secondary endpoints: | 12 |
| Research design | 12 |
| Type of study | 12 |
| Experimental diagram | 13 |
| Subject selection | 14 |
| Inclusion criteria | 14 |
| Exclusion criteria | 14 |
| Treatment allocation | 15 |
| Procedures for randomization | 15 |
| Dosage and administration | 15 |
| Study process | 16 |
| Screening phase | 16 |
| Treatment period | 17 |
| Termination phase | 17 |
| Follow-up phase | 18 |
| Response evaluation | 18 |
| Safety evaluations | 18 |
| Safety endpoints | 19 |
| Clinical symptoms | 19 |
| Laboratory examination | 19 |
| Adverse event | 19 |
| Definition and record of an adverse event | 19 |
| Classification of adverse event severity | 19 |
| Relevance | |
| Serious adverse event | 20 |
| Definition of an unexpected adverse event | 21 |
| Expected adverse events | 21 |
| Procedures of all adverse event | 21 |
| Monitoring committee | 22 |
| Statistical methods | 22 |
| Sample size estimation | 23 |

| Statistical analysis | 23 |
|--------------------------------------------------------------|----|
| Management of product quality complaint | 24 |
| Procedures | 24 |
| Study drug information | 24 |
| Ethical statement | 25 |
| Ethical principles | 25 |
| Information and informed consent | 25 |
| Withdrawal from the study | 26 |
| Identity and privacy of patients | 26 |
| Responsibility of independent ethics committee | 27 |
| Responsibility of investigator | 28 |
| Publications | |
| Organization and responsibility | |
| Appendix | 30 |
| Appendix 1. The score of bleeding | 31 |
| Appendix 2. ECOG score | |
| Appendix 3. Criteria for IBMTR severity index for acute GVHD | 33 |
| Appendix 4. NIH global severity of chronic GVHD | |
| Appendix 5. The table of study procedure | |
| Appendix 6: Patient consent form for study participation | |

#### **Protocol amendments**

| Protocol version | Issue date |
|------------------|---------------|
| Vision 1.0 | Sep. 01, 2015 |
| Vision 2.0 | Mar. 21, 2016 |
| Vision 3.0 | Aug. 07, 2017 |

Vision 3.0 (Aug. 07, 2017)

#### **Applicable Section**

#### Study centers:

The First Affiliated Hospital of Soochow University, Suzhou 215006, China; Nanfang Hospital, Southern Medical University, Guangzhou 510515, China; Rui Jin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai 200025, China;

Peking University People's Hospital, Beijing 100044, China;

Wuhan Union Hospital, Wuhan 430022, China;

Qilu Hospital of Shandong University, Jinan 250012, China.

#### **Description of Changes**

#### Three other institutions took part in this study:

Fujian Medical University, Union Hospital, Fuzhou 350001, China; Children's Hospital of Soochow University, Suzhou 215025, China; Hebei Yanda Lu Daopei Hospital, Langfang 065201, China.

Vision 2.0 (Mar. 21, 2016)

#### **Applicable Section**

#### Secondary objectives and secondary endpoints:

To evaluate the megakaryocyte counts, white blood cell counts, hemoglobin level, renal and liver function at week 4.

#### **Description of Changes**

#### Secondary objectives and secondary endpoints:

To evaluate the megakaryocyte counts and survival during a follow-up of 24 weeks.

#### **Protocol Summary**

#### **Study centers**

- The First Affiliated Hospital of Soochow University, Suzhou 215006, China:
- Nanfang Hospital, Southern Medical University, Guangzhou 510515, China;
- Fujian Institute of Hematology, Fuzhou 350001, China;
- Children's Hospital of Soochow University, Suzhou 215025, China;
- Hebei Yanda Lu Daopei Hospital, Langfang 065201, China;
- Rui Jin Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai 200025, China;
- Peking University People's Hospital, Beijing 100044, China;
- Wuhan Union Hospital, Wuhan 430022, China;
- Qilu Hospital of Shandong University, Jinan 250012, China.

#### **Principal Investigator**

Yue Han, MD, PhD; Depei Wu, MD, PhD.

#### Methodology

A prospective, open-label, three-arm, multicenter, randomized clinical trial.

#### **Primary objective**

To assess the efficacy of low-dose decitabine in patients with refractory prolonged isolated thrombocytopenia after hematopoietic cell transplantation.

#### Secondary objectives

To evaluate the number of megakaryocytes and survival during a follow-up of 24 weeks.

#### Inclusion criteria

- Platelet count < 30 × 10<sup>9</sup>/L for more than 60 days post-HCT;
- Recovered neutrophil and hemoglobin concentrations;
- Donor chimerism >95% detected by short-tandem repeat-polymerase chain reaction;
- No response to conventional treatments for thrombocytopenia for a duration of at least 4 weeks;

#### **Exclusion criteria**

- Patients with disease relapse;
- · Active infections requiring treatment;
- Grade III-IV acute GVHD or severe chronic GVHD according to National Institute of Health criteria;
- Severe organ damage (cardiac, renal and/or hepatic dysfunction greater than grade 2 according to the Common Terminology Criteria for Adverse Events V5.0);

- Thrombosis requiring treatment;
- Received decitabine following the current transplantation;

#### Intervention

- Arm A: decitabine 15 mg/m² daily for consecutive 3 days, combined with recombinant human thrombopoietin 300 U/kg daily;
- Arm B: decitabine 15 mg/m<sup>2</sup> daily for consecutive 3 days alone;
- Arm C: conventional therapies;

**Total number of patients**: 96

Total duration of the study: 4 years

#### **Background**

## Refractory prolonged isolated thrombocytopenia after allogeneic hematopoietic cell transplantation

Thrombocytopenia is a frequent and worrisome complication after hematopoietic cell transplantation (HCT)<sup>1-4</sup>, described in 5-37% of the recipients<sup>5-8</sup>, which is not only associated with disease relapse or graft rejection, but also significantly correlates with increased incidence of transplant-related complications and a higher mortality rate<sup>1,9</sup>. However, it is very difficult to decipher the precise etiology of thrombocytopenia during the post-transplant period in a clinical setting. Possible pathogenesis includes graft-failure, drugs, veno-occlusive disease, cytomegalovirus infection, opportunistic infection, recurrence of the primary disease, graft-versus-host disease (GVHD), etc<sup>4</sup>.

The major causes of thrombocytopenia include accelerated peripheral platelet destruction by antiplatelet antibodies and the insufficient production of platelets from marrow megakaryocytes (MKs). In previous studies, both increased platelet turnover and impaired thrombopoiesis have been reported to be involved in the development of thrombocytopenia after HCT<sup>6</sup>. Furthermore, impaired bone marrow (BM) vascular microenvironment also contribute to the occurrence of thrombocytopenia after allo-HCT, including cellular elements (bone marrow endothelial cells, perivascular cells, etc), and MK-active factors (stromal cell-derived factor-1, vascular endothelial growth factor, etc)<sup>10</sup>.

Previous studies showed thrombocytopenia after HCT was closely associated with a poor survival, and any haemorrhagic complications may thus prove to be fatal<sup>5</sup>. Therefore, successful management of thrombocytopenia following HCT is essential in order to achieve and maintain a favorable outcome. Some patients may respond to conventional practices including recombinant human

thrombopoietin (rhTPO), interleukin-11, immunoglobulin, methylprednisolone. However, there is also a proportion of patients without an identified cause who are often resistant to these conventional treatments for thrombocytopenia. We describe these patients as refractory prolonged isolated thrombocytopenia (RPIT).

#### rhTPO for thrombocytopenia

TPO is a hematopoietic growth factor that stimulates the proliferation and differentiation of hematopoietic stem cells, primitive progenitors, megakaryocytes, and platelets<sup>11-13</sup>. In vitro and vivo studies, TPO has been proven to be the principal physiologic cytokine that stimulates platelet production<sup>14-15</sup>. Both preclinical and clinical studies revealed that rhTPO or TPO receptor (TPOR) agonists could promote platelet recovery in thrombocytopenia patients<sup>16-19</sup>. TPOR agonists, such as eltrombopag and romiplostim, have also been shown effective in thrombocytopenia patients after HCT<sup>19-20</sup>, which still needs more large-scale, prospective studies to verify.

#### Decitabine for thrombocytopenia after HCT

Decitabine (5-aza-2´-deoxycytidine) is a deoxycytidine analog which acts as a hypomethylating agent that is incorporated into DNA and forms irreversible covalent adducts with DNA-methyltransferases. Emerging studies showed decitabine can increase platelet count and megakaryocyte numbers<sup>21-24</sup>. Decitabine was found to be able to induce mouse megakaryoblastic cell to differentiate into a megakaryocyte-like polyploidy cells. Additionally, a 30% platelet count increase in mice 12 hours after the injection of decitabine at a clinically relevant dose (15 mg/m²) was observed<sup>21</sup>. In vitro study, dectibine can promote megakaryocyte maturation and platelet production and enhance TRAIL expression in megakaryocytes of immune thrombocytopenia<sup>24</sup>. Our previous study suggested that low-dose decitabine, could significantly

increase the platelet count by increasing the number of megakaryocytes of thrombocytopenia after HCT, but with limited cases<sup>22</sup>. Herein, a prospective, open-label, three-arm, randomized clinical trial will be conducted to validate the efficacy and safety of low-dose decitabine in RPIT patients after HCT and to preliminarily explore the potential mechanisms of RPIT.

#### Reference

- 1. Kim DH, Sohn SK, Jeon SB, et al. Prognostic significance of platelet recovery pattern after allogeneic HLA-identical sibling transplantation and its association with severe acute GVHD. Bone Marrow Transplantation 2006; 37(1): 101-108.
- 2. Akpek G, Lee SJ, Flowers ME, et al. Performance of a new clinical grading system for chronic graft-versus-host disease: a multicenter study. Blood 2003; 102(3): 802-809.
- 3. First LR, Smith BR, Lipton J, et al. Isolated thrombocytopenia after allogeneic bone marrow transplantation: existence of transient and chronic thrombocytopenic syndromes. Blood 1985; 65(2): 368-374.
- 4. Nash RA, Gooley T, Davis C, et al. The Problem of Thrombocytopenia after Hematopoietic Stem Cell Transplantation. Oncologist 1996; 1(6): 371-380.
- 5. Ramrez P, Brunstein CG, Miller B, et al. Delayed platelet recovery after allogeneic transplantation: a predictor of increased treatment-related mortality and poorer survival. Bone Marrow Transplantation 2011; 46(7): 981-986.
- 6. Yamazaki R, Kuwana M, Mori T, et al. Prolonged thrombocytopenia after allogeneic hematopoietic stem cell transplantation: associations with impaired platelet production and increased platelet turnover. Bone Marrow Transplant 2006; 38(5): 377-384.
- 7. Bruno B, Gooley T, Sullivan KM, et al. Secondary failure of platelet recovery after hematopoietic stem cell transplantation. Biol Blood Marrow Transplant 2001; 7(3): 154-162.
- 8. Klumpp TR, Block CC, Caligiuri MA, et al. Immune-mediated cytopenia following bone marrow transplantation. Case reports and review of the literature. Medicine (Baltimore) 1992; 71(2): 73-83.
- 9. Kuzmina Z, Eder S, Bohm A, et al. Significantly worse survival of patients with NIH-defined chronic graft-versus-host disease and thrombocytopenia or progressive onset type: results of a prospective study. Leukemia 2012; 26(4): 746-756.
- 10. Kong Y, Hu Y, Zhang XH, et al. Association between an impaired bone marrow vascular microenvironment and prolonged isolated thrombocytopenia after allogeneic hematopoietic stem cell transplantation. Biol Blood Marrow Transplant 2014; 20(8): 1190-1197.
- 11. Kaushansky K. Thrombopoietin: the primary regulator of platelet production. Blood 1995; 86(2): 419-431.
- 12. Wendling F. Thrombopoietin: its role from early hematopoiesis to platelet production. Haematologica 1999; 84(2): 158-166.

- 13. Kaushansky K. Thrombopoietin: understanding and manipulating platelet production. Annu Rev Med 1997; 48: 1-11.
- 14. Kaushansky K, Lok S, Holly RD, et al. Promotion of megakaryocyte progenitor expansion and differentiation by the c-Mpl ligand thrombopoietin. Nature 1994; 369(6481): 568-571.
- 15. Alexander WS, Roberts AW, Nicola NA, et al. Deficiencies in progenitor cells of multiple hematopoietic lineages and defective megakaryocytopoiesis in mice lacking the thrombopoietic receptor c-Mpl. Blood 1996; 87(6): 2162-2170.
- 16. Thachil J, Salter I and George J N. Complete remission of refractory immune thrombocytopenia (ITP) with a short course of Romiplostim. Eur J Haematol 2013; 91(4): 376-377.
- 17. Neunert CE, Grace RF. Thrombopoietin-receptor agonists in children with immune thrombocytopenia. Lancet 2015; 386(10004): 1606-1609.
- 18. Wang Y, Wang Z, Wu L, et al. Recombinant human thrombopoietin is an effective treatment for thrombocytopenia in hemophagocytic lymphohistiocytosis. Ann Hematol 2013; 92(12): 1695-1699
- 19. Battipaglia G, Ruggeri A, Brissot E, et al. Safety and feasibility of romiplostim treatment for patients with persistent thrombocytopenia after allogeneic stem cell transplantation. Bone Marrow Transplant 2015; 50(12): 1574-1577.
- 20. Reid R, Bennett JM, Becker M, et al. Use of eltrombopag, a thrombopoietin receptor agonist, in post-transplantation thrombocytopenia. Am J Hematol 2012; 87(7): 743-745.
- 21. Wang J, Yi Z, Wang S, et al. The effect of decitabine on megakaryocyte maturation and platelet release. Thrombosis and Haemostasis 2011; 106(2): 337-343.
- 22. Han Y, Tang Y, Chen J, et al. Low-Dose Decitabine for Patients With Thrombocytopenia Following Allogeneic Hematopoietic Stem Cell Transplantation: A Pilot Therapeutic Study. JAMA Oncol 2015; 1(2): 249-251.
- 23. van den Bosch J, Lübbert M, Verhoef G, et al. The effects of 5-aza-2-deoxycytidine (Decitabine) on the platelet count in patients with intermediate and high-risk myelodysplastic syndromes. Leukemia Research 2004; 28(8): 785-790.
- 24. Zhou H, Hou Y, Liu X et al. Low-dose decitabine promotes megakaryocyte maturation and platelet production in healthy controls and immune thrombocytopenia. Thromb Haemost 2015; 113(5): 1021-1034.

#### Rationale of this study

- RPIT, a frequent complication after HCT, is often resistant to conventional treatment and leads to a poor prognosis;
- ➤ A proportion of patients without an identified cause are often resistant to conventional treatments for thrombocytopenia;
- ➤ We previously demonstrated low-dose decitabine, a hypomethylating agent, could significantly increase the platelet count by increasing the number of megakaryocytes;
- ➤ This randomized trial will be conducted to validate the efficacy and safety of low-dose decitabine in RPIT patients after HCT and to preliminarily explore the potential mechanisms.

#### Study objectives

#### Primary objective and primary endpoint

#### **Primary objective:**

This study aims to validate the efficacy of low-dose decitabine in HCT-RPIT patients.

#### **Primary endpoint:**

The primary endpoint is the recovery of platelet count of HCT-RPIT patients.

#### Secondary objectives and secondary endpoints:

To evaluate the megakaryocyte counts and survival during a follow-up of 24 weeks.

#### Research design

#### Type of study

This is a prospective, open-label, randomized, three-arm clinical trial.

#### **Experimental diagram**

The overall design of the study is shown in Figure 1.



<sup>&</sup>lt;sup>a</sup> refers to a platelet count < 30 × 10<sup>9</sup>/L

Figure 1. The flow chart of the overall study design

Notes: HCT, hematopoietic cell transplantation; GVHD, graft-versus-host disease; rhTPO, recombinant human thrombopoietin.

<sup>&</sup>lt;sup>b</sup> refers to neutrophil count < 1.0 × 10<sup>9</sup>/L and/or red blood cells transfusion dependent

#### **Subject selection**

#### Inclusion criteria

- ➤ Platelet count < 30 × 10<sup>9</sup>/L for more than 60 days post-HCT;
- Recovered neutrophil and hemoglobin concentrations;
- Donor chimerism >95% detected by short-tandem repeat-polymerase chain reaction;
- ➤ No response to conventional treatments for thrombocytopenia (rhTPO, immunoglobulin, rituximab and glucocorticoid, either alone or in combination) for a duration of at least 4 weeks.

#### Exclusion criteria

- > Patients with disease relapse:
- Active infections requiring treatment;
- Grade III-IV acute GVHD or severe chronic GVHD according to National Institute of Health criteria;
- Severe organ damage (cardiac, renal and/or hepatic dysfunction greater than grade 2 according to the Common Terminology Criteria for Adverse Events V5.0);
- Thrombosis requiring treatment;
- > Received decitabine following the current transplantation.

#### Note:

- ➤ If a subject's status changes (including laboratory results) and meets the exclusion criteria after screening but before the first dose of the study drug is given, he/she should be excluded from this study.
- ➤ Patients suffered from disease relapse would be excluded from this study during the 4-week study period as the relapse evidence of a small number of patients is negative during screening procedure, but it turns to be positive in the process of disease progression.

#### **Treatment Allocation**

Subjects will be randomized after the investigator has verified that all eligibility criteria have been met. Subjects will be randomized in a 1:1:1:1 ratio to receive decitabine in combination with rhTPO (Arm A), decitabine alone (Arm B) or conventional treatment except decitabine (Arm C).

#### Procedures for randomization

Completely randomized block design method was performed to assign the patients into the 3 arms. For each study site, we produced the random series and corresponding assigning arm A, B, C, in which the block equals to 5 and length equals to 6. If the length <= 2 then the group is A, 3-4 is B, and 5-6 is C.

#### Dosage and administration

#### **Treatment:**

Arm A: decitabine 15 mg/m<sup>2</sup> daily intravenously for consecutive 3 days (day 1 to day 3), combined with rhTPO 300 U/kg daily subcutaneously beginning on day 4 and continuing until the response was achieved or the time of initial evaluation (day 28);

Arm B: decitabine 15 mg/m<sup>2</sup> daily intravenously for consecutive 3 days (day 1 to day 3) alone;

Arm C: conventional therapies with recommended options including rhTPO, eltrombopag, immunoglobulin, rituximab, interleukin-11 and glucocorticoids, alone or in combination.

#### Note:

➤ For patients with neutropenia (neutrophils ≤0.5×10<sup>9</sup>/L), the granulocyte colony-stimulating factor (G-CSF, 5 ug/kg·d) should be administrated to reduce the chance of neutropenia related infections. Prophylactic platelet transfusion is required for no-bleeding patients with platelet counts lower than 20×10<sup>9</sup>/L and those with bleeding and platelet counts lower than

- $30 \times 10^9$ /L. For those with severe anemia (hemoglobin  $\le 60$  g/L), washed red blood cells should be given.
- ➤ There is no need of special treatment for transient fever (except infections related fever), muscle soreness, dizziness.
- Decitabine treatment should be suspended when some non-hematologic toxicities appear as follows:
- Serum creatinine ≥ 2.0mg/dL;
- Serum aminotransferase or total bilirubin higher than 2 fold the upper-limit of normal level.

#### Concomitant therapy

Except the study drug, other therapies (including immunosuppressant, antibiotics, proton-pump inhibitor, diuretic, nutritional therapy, etc) must be recorded in the eCRF for the main study treatment period.

The concurrent administration of other drugs which are known as myelosuppression is not recommended unless absolutely necessary.

#### Study process

#### Screening phase (3 days)

- Inclusion /Exclusion Criteria
- Demographic data: age, sex, nationality, address, spouse's characteristics, contact information.
- ➤ General information: past history, allergic history, previous disease and status, transplant type, conditioning regimen, number of infused stem cells, the time of neutrophils reconstitution after HCT, the time of enrollment after HCT, other complications except thrombocytopenia, other myelosuppression therapies.
- Physical examination: height, body weight, blood pressure, body temperature, heart rate, body surface area, respiratory and cardiovascular

system examination, nervous system examination, Eastern Cooperative Oncology Group (ECOG) score, etc.

- ➤ Laboratory examination:
- Blood analysis: blood routine test, blood biochemistry, virological testing, Tlymphocyte subsets, platelet-associated antibody, serum TPO level\*
- BM examination: marrow morphology examination (megakaryocyte including: platelet-shedding megakaryocyte, granular megakaryocyte, naked megakaryocyte), endothelial progenitor cell\*, etc.

Note: \* represents blood or BM needs to be collected and sent to the group leader institution for examination, in which blood 2 mL is anticoagulated using sodium citrate and BM 8 mL is anticoagulated by ethylene diamine tetraacetic acid (EDTA). Both bone marrow and blood should be transported under 4°C.

➤ Electrocardiogram test.

#### Treatment period (28 days)

- Drugs will be given based on the protocol;
- ➤ Blood routine test and blood biochemistry are performed once a day and once a week, respectively.
- Important vital signs are recorded;
- Adverse events will be recorded and managed according to this protocol.

#### **Termination phase**

- Demographic data: age, sex, nationality, address, spouse's characteristics, contact information.
- ➤ General information: past history, allergic history, previous disease and status, transplant type, conditioning regimen, number of infused stem cells, the time of neutrophils reconstitution after HCT, the time of enrollment after HCT, other complications except thrombocytopenia, other myelosuppression therapies.

- ➤ Physical examination: height, body weight, blood pressure, body temperature, heart rate, body surface area, respiratory and cardiovascular system examination, nervous system examination, ECOG score, etc.
- ➤ Laboratory examination:
- Blood analysis: blood routine test, blood biochemistry, virological testing, Tlymphocyte subsets, platelet-associated antibody, serum TPO level\*
- Bone marrow examination: marrow morphology examination
   (megakaryocyte including: platelet-shedding megakaryocyte, granular megakaryocyte, naked megakaryocyte), endothelial progenitor cell\*, etc.

Note: \* represents blood or BM needs to be collected and sent to the group leader institution for examination, in which blood 2 mL is anticoagulated using sodium citrate and BM 8 mL is anticoagulated by ethylene diamine tetraacetic acid (EDTA). Both bone marrow and blood should be transported under 4°C.

> Electrocardiogram test.

#### Follow-up phase (6 months)

- ➤ Routine blood examination will be repeated once every 1 month;
- > The changes of other complications;
- Survival will be long-term recorded until death.

#### Response evaluation

- ➤ Response: A sustained increase (stable or increasing level) of at least 30×10<sup>9</sup>/L independent of transfusion for 3 days.
- ➤ No response: The requirements for "response" can not be met.

#### Safety evaluations

Safety and tolerability are assessed throughout the study.

#### Safety endpoints

White blood cell count, hemoglobin, liver function, renal function.

#### **Clinical symptoms:**

Newly occurred symptoms during the study period: fever, nausea, cough, somnolence, depression, constipation, diarrhea, petechia, edema, pharyngitis, pulmonary edema, atrial fibrillation, tachycardia, mycobacterium avium complex infectious, hyperglycemia, neutropenia, anemia.

#### Laboratory examination

Blood routine test, blood biochemistry, virological testing, electrocardiogram, etc.

#### Adverse event

#### Definition and record of an adverse event

Adverse events are defined as any harmful medical manifestations occurring in a person who participates in a biomedical research whether this manifestation is related to the research or the product used in the research. An adverse effect may be any unfavourable or unexpected sign (including abnormal laboratory results), any symptom or temporary disorder associated with the use of the product, with or without relation to the product. The clinically significant abnormality must be reported as an adverse event (AE) in the eCRF, and AE is supposed to record the time of occurrence, the stage of severity, the duration of time, measures and outcomes.

#### Classification of adverse event severity

Every case report is performed by the grade of severity about drug adverse reactions:

Mild: usually transient symptoms unaffecting the daily life;

- Moderate: symptoms probably affecting the daily life;
- Severe: symptoms seriously affecting the daily life.

#### Relevance

- ➤ Definite relevance: The adverse event is clearly related to the investigational agent. For example, an event that follows a reasonable temporal sequence from administration of the study intervention abides by a known or expected response pattern to the suspected intervention, which improves by stoppage and reappears through repeated exposures, but is unable to be reasonably explained by the known characteristics of the subject's clinical state;
- ➤ Possible relevance: An adverse event that follows a reasonable temporal sequence from administration of the study intervention abides by a known or expected response pattern to the suspected intervention, which can be easily induced by various other factors;
- ➤ Irrelevance: The adverse event is clearly uncorrelated with the research agent or procedure. For example, there exists another plausible cause, and/or a clinically plausible temporal sequence is inconsistent with the onset of the event and the study intervention and/or a causal relationship is considered biologically implausible.

#### Serious adverse event:

A serious adverse event (SAE) event is defined as the event with one of the following consequences:

- Death;
- ➤ Life-threatening condition;
- Hospitalization or extension of hospitalization;
- Temporary or permanent disability;
- Congenital anomaly or malformation;

Important medical events: although the event caused by the drug which may endanger the subjects may not be life-threatening and result in death or require hospitalization, medical or surgical intervention requires to be taken to prevent one of the outcomes based on the appropriate medical judgment.

#### Definition of an unexpected adverse event:

An unexpected adverse event of the product is defined as the event with the nature, severity or course non-corresponding to the product information mentioned in the summary when it is authorized or in the investigator's brochure when it is not authorized.

#### **Expected adverse events:**

#### Due to myelosuppression

Neutropenia related infections, fever;

Bleeding: ecchymosis, petechial, haematemesis, hemoptysis, melena, hematuresis, etc;

Weary, somnolence, pale, etc (due to anemia);

#### Due to other non-hematological toxicity

Liver dysfunction;

Renal dysfunction;

#### > Related to the haematological disease

Death

Relapse of any kind

#### > Related to drug allergy

Erythra, edema, pruritus, swelling, etc.

#### Procedures of all adverse event

Investigators must immediately take necessarily measures at once to protect subjects' safety, when serious adverse events occur. Furthermore, all adverse

events should be followed up and investigated, and detailed records are supposed to be made and signed.

All serious and non-serious AEs and special situation will be reported from the signature to completion of the subject's last study-related procedure (which may include the follow-up contact for safety). SAEs must be reported using the Serious Adverse Event Form. The sponsor will evaluate any safety information that is spontaneously reported by an investigator beyond the time frame specified in the protocol.

All AEs, regardless of the severity or presumed relationship with the study treatment, must be recorded in the source document and eCRF using medical terminology. Whenever possible, diagnosis should be made when signs and symptoms are caused by the common etiology. Investigators must record their opinions on the relationship between AEs and the study treatment in the eCRF. All measures required for (serious) AEs must be recorded in the source document and reported according to sponsor instructions.

#### Monitoring committee

A safety committee comprised of 3 persons independent of the trial will be organized and will meet to check the safety related to the study treatment during the study. In terms of the overall mortality of each arm and serious adverse events, review will be performed by the independent safety committee. The committee is responsible for haemovigilance/pharmacovigilance of the study and acts as an additional

warning sign against haemovigilance/pharmacovigilance of the study.

#### Contact

Yue Han (Email: hanyue@suda.edu.cn), Depei Wu (wudepei@suda.edu.cn), The First Affiliated Hospital of Soochow University, Suzhou 215006, China.

#### Statistical methods

Statistical analysis will be done by the sponsor or under the authority of the sponsor. A general description of the statistical methods to be used to analyze the efficacy and safety data is outlined below. Baseline for all analyses will be the day of randomization unless otherwise specified.

#### Sample size estimation

We used the formula of sample size estimate when comparing the independent rates more two groups. According to the previous study, among the 3 groups, we suppose the biggest effective rate was 80% ( $P_{\text{max}}$ ), and the lowest rate was about 35% ( $P_{\text{min}}$ ). Under the condition of  $\alpha$ =0.05(2-tailed),  $\beta$ =0.20(1-tailed), v=2, so  $\lambda$ =9.63, the theoretical sample size for each group can be calculated as follow,

$$n = \frac{\lambda}{2(\arcsin\sqrt{p_{max}} - \arcsin\sqrt{p_{min}})^2} = \frac{9.63}{2(\arcsin\sqrt{0.80} - \arcsin\sqrt{0.35})^2}$$
$$= 21.42$$

Taking account of the 20% of loss rate of follow up, so the sample size for each group at least was 25, and the total sample size should at least be 75.

#### Statistical analysis

Completely randomized block design method was performed to assign the patients into the 3 arms. Numerical data was presented as medians with interval quartile range (IQR), and categorical data were shown as proportions. One-way ANOVA was used to compare the difference for the means among 3 treatment arms. Since there was no statistical difference in response or survival between Arms A and B, these data were combined for subsequent comparisons to Arm C. Chi-square test or Wilcoxon rank test was used to compare the difference for the proportions among 3 treatment arms. Kaplan-Meier method was performed to estimate the 1-year survival rate for the 3 arms respectively and log-rank test to compare their difference for the survival

curves. Cox model and logistic model were used to estimate independent association for the HR (hazard ratio), OR (odds ratio) and 95% CI (confidence interval) among the treatment arms. A significance level was set as a 2-tailed P value of < .05. All the analyses used the SPSS 19.0 (SPSS Inc.).

#### Management of product quality complaint

A product quality complaint (PQC) is defined as any suspicion of a product defect related to manufacturing, labeling, or packaging, ie, any dissatisfaction relative to the identity, quality, durability, or reliability of a product, including its labeling or package integrity. PQCs may have an impact on the safety and efficacy of the product. Timely, accurate, and complete reporting and analysis of PQC information from clinical studies are crucial for the protection of subjects, investigators, and the sponsor, and are mandated by regulatory agencies worldwide.

#### **Procedures**

All initial PQCs must be reported to the sponsor by the investigational staff within 24 hours after being made aware of the event.

If the defect is combined with an SAE, the investigational staff must report the PQC to the sponsor according to the SAE reporting timelines. A sample of the suspected product should be maintained for further investigation if requested by the sponsor.

### Study drug information

- ➤ Decitabine is a kind of white sterile lyophilized powder, placed in a clear, colorless vial. Each 20 mL vial contains 25 mg decitabine.
- ➤ rhTPO is a sterile, clear, colorless liquid. The single-use vial contains 15 000 U rhTPO when the fill volume is 1.0 mL.

#### Ethical statement

#### **Ethical principles**

The study should be carried out in accordance with Helsinki declaration proposed by World Medical Association and subsequent amendments and approved by the Independent Ethics Committee (IEC) before implementation.

#### Information and informed consent

- ➤ All the patients who agree to participate should be asked to sign the informed consent form to prove their approval for participation in this study. The informed consent form must be signed and dated personally by the patients and investigators.
- ➤ Before obtaining the informed consent, the investigators must provide sufficient information to the patients who are potential participants in this study:
- The investigators should orally inform the patients of all the relevant circumstances of this study;
- The information provided to patients must be fully and easily understood by non-professionals, so that they can make a decision according to their own willingness based on their full understanding of this study;
- Additionally, the patients voluntarily participate in the study, and are free to
  quit from the study at any time, without any reasons. The subsequent
  treatment of patients is not under the influence of unwilling to participate or
  quitting from the study.
- All the patients who agree to participate should be asked to sign the Informed Consent Form (ICF) to prove their approval for participation in this study. The ICF must be signed and dated personally by the patients and the investigators;

➤ The signed ICF will be kept in the Data Center and must be safely kept for future review at any time throughout the study.

#### Withdrawal from the study

The main withdrawal criteria are as following:

- Relapsed during the first 4 weeks of treatment;
- Changes in the patient's condition after inclusion, which suggests that the study protocol is unsuitable for the patient;
- Severe complications affecting the implementation of the study treatment;
- Patients who are confirmed to require emergency treatment due to other diseases after inclusion;
- > Treatment unmated with the study protocol;
- ➤ Patients who voluntarily quit or discontinue any examination, treatment and monitoring required by the study for personal reasons at any stage after inclusion in this study. The PI also has the right to withdraw patients from the study if he/she feels that the withdrawal is in the best interests of the patients.

#### Identity and privacy of patients

- After obtaining an ICF, each enrolled patient is assigned a subject number (allocation number). This number will represent the identity of the patient during the study and for the retrieving of dedicated clinical research database;
- ➤ Throughout the study, several measures will be taken to minimize any breaches of personal information, including:
- Only the PI and co-investigators will be able to link to the research data of the patients to themselves through the identifiable table after authorization;
- Collection, transmission, handling and storage of the study data must comply with the data protection and privacy regulations.

#### Responsibility of independent ethics committee

The responsibilities of independent ethics committee include:

- Review of this study;
- ➤ Evaluate this study to determine if risks to which patients are exposed have been duly minimized and whether these risks are reasonable compared to expected benefits;
- Check the study protocol and relevant documents (patient information sheet, ICF, CRF, etc.) submitted by the Research Committee before beginning of the study;
- ➤ Provide the written proof of ethical review opinions, the written proof of the date of the review meeting, the written proof of the members presenting at the meeting and voting members, the written proof of recording of the reviewed versions of study protocol, ICF and other related documents, and if possible, a copy of the minutes, to the Research Committee. The study can begin only after obtaining the written proof of favorable opinions/approval of the IEC;
- Supervise the legitimacy of the process of informed consent;
- ➤ Ensure the safety of patients during the research process by examining the reported safety information. The investigators should report to the IEC on any therapeutic complications which may affect the safety of patients.

  When complications that affect the patient safety occur, the IEC should inform PI to withdraw patients from the study and use any possible treatment to cure patients. If the PI decides not to withdraw patients from the study, he should provide a written proof of explanation to the IEC;
- ➤ Review the reasonableness of the costs incurred by patients in the course of the study through a selective check for hospitalization expenses. When the patient has indications for off-label use of drugs, the IEC will receive the notice and the description of relevant situation from the investigators. The IEC should record the relevant records:

- ➤ Review the revisions of the study protocol, and any changes must be approved by the IEC before they are adopted. Unless the change is necessary to eliminate an immediate hazard to the patients, in which case the IEC should be informed as soon as possible;
- ➤ Review the progress of the study annually and the close-out report submitted by the Research Committee at the end of the trial.

#### Responsibility of investigator

The responsibilities of investigators are as follows:

- ➤ Investigators, participated in the clinical trial, should be obtained certificate for assistant practicing doctor, resigned and attended the training of the GCP guidelines and the correlation of laws and regulations, possessed specialty, qualification and ability in clinical trial.
- ➤ Subjects are adequately recruited by the investigator during required time according to the clinical trial, and operation capacity and possibility to be qualified the item should be evaluated by the previous working experience.
- ➤ Investigators are familiar with clinical trial protocols and execute instruction strictly according to the protocols and case report form.
- ➤ In all adverse events, subjects must be taken appropriate therapies and made a contact with the investigator as soon as possible. Investigators will take responsibilities of relevant medical decision of clinical trial to ensure subjects that is taken adequate medical treatment.
- ➤ Any information on the case report form possesses original data, to ensure the case history and case report form filled in truly, accurately, completely, timely, regularly and legally.
- ➤ Subjects will be illustrated the relevant situation where the clinical trial is fully consent by Ethics Committee. The informed consent will be acquired and, during the process, it must meet the specification.

- Supervision and inspection will be received by supervisor and inspector assigned by sponsor to ensure the quality of clinical trial.
- Any advices and suggestions focused on the study protocols might be submit to the principal institution of clinical research, and made a discussion with sponsor and coordination institutions to decide whether adopting the above advice or suggestions, during the clinical trial executed by each institutions.

#### **Publications**

- ➤ All the data collected during this study are the property of the study sponsor and cannot be communicated in any case to a third party without the written agreement of the investigator.
- Any publication or communication (oral or written) will be decided from a common agreement between the investigators and will respect the international recommendations: "Uniforms Requirements for Manuscripts Submitted to Biomedical Journals" (http://www.cma.ca/publications/mwc/uniform.htm): notably, an authorship will be proposed to each clinical center participating in the study and to each member of the steering committee according to his/her actual participation.

### Organization and responsibility

The Research Committee is responsible for developing study protocol, auditing patient eligibility and guiding interpretation of informed consent. It is also responsible for collection of complication reports, guiding diagnosis and treatment of complications and emergency intervention for serious complications, as well as approving the content and distribution of all publications related to the study.

## **Appendix**

- Appendix 1. The score of bleeding
- Appendix 2. ECOG score
- Appendix 3. Criteria for IBMTR severity index for acute GVHD
- Appendix 4. NIH global severity of chronic GVHD
- Appendix 5. The table of study procedure
- Appendix 6. Patient consent form for study participation

## Appendix 1. The score of bleeding\*

| Grade | Manifestation |
|---|---|
| Score 0 | No bleeding. |
| Score 1 | Occult bleeding in secretion, including mild petechia or minimal |
| | vaginal bleeding. |
| Score 2 | Minor bleeding without the requirement of RBC transfusion, such |
| | as ecchymosis, epistaxis, line oozing, vaginal bleeding, skin |
| | bleeding, mild hematemesis, melena, mild hematuria. |
| Score 3 | Bleeding that can cause a rapid fall of hematocrit and needs one |
| | or more units of RBC transfusion per day over the expected rate |
| | of an individual, or fail to obtain a post-transfusion increment at |
| | active bleeding. |
| Score 4 | Life-threatening bleeding, defined as either massive bleeding |
| | causing severe hemodynamic compromise or bleeding into a |
| | vital organ, such as intracranial hemorrhage, pericardial |
| | hemorrhage, diffuse alveolar hemorrhage. |

**Notes**: RBC=red blood cell; \*Nevo S, Enger C, Hartley E, et al. Acute bleeding and thrombocytopenia after bone marrow transplantation. Bone Marrow Transplant. 2001;27(1):65-72.

## Appendix 2. ECOG score\*

| Grade | Performance status |
|---|---|
| 0 | Fully active, able to carry on all pre-disease performance without |
| | restriction. |
| 1 | Able to move freely and take mild physical activity, such as |
| | housework and office work, but restricted in severe physical activity. |
| 2 | Able to move freely and take care of himself, but loss of work |
| | capability; doing activities for more than half of the waking hours. |
| 3 | Capable of taking care of himself partially, confined to the bed or chair |
| | for more than half of the waking hours. |
| 4 | Completely disabled, unable to take care of himself and totally |
| | confined to the bed or chair. |
| 5 | Dead |

**Notes**: ECOG=Eastern Cooperative Oncology Group; \* Oken M, Creech R, Tormey D, et al. Toxicity and response criteria of the Eastern Cooperative Oncology Group. Am J Clin Oncol. 1982;5:649-655.

Appendix 3. Criteria for IBMTR severity index for acute GVHD\*

| Skin in | volvemer | nt | | Liver involvement Gastro | | | Gastroin | trointestinal involvement |
|---|---|---|---|---|---|---|---|---|
| Index | Stage | Rash | _ | Stage | Total bilirubin | _ | Stage | Volume of diarrhea |
| | (max.) | range | | (max.) | (µmol/L) | | (max.) | (ml/d) |
| Α | 1 | <25% | | 0 | <34 | | 0 | <500 |
| В | 2 | 25%- 50% | or | 1-2 | 34-102 | or | 1-2 | 550-1 500 |
| С | 3 | >50% | or | 3 | 103-255 | or | 3 | >1 500 |
| D | 4 | Bullae | or | 4 | >255 | or | 4 | Severe pain and |
| | | | | | | | | ileus |

**Notes**: GVHD=graft-versus-host disease; \*Rowlings PA, Przepiorka D, Klein JP, et al. IBMTR Severity Index for grading acute graft-versus-host disease: retrospective comparison with Glucksberg grade. Br J Haematol. 1997;97(4):855-64.

#### Appendix 4. Criteria of chronic GVHD\*

| Severity | Manifestation |
|----------|--------------------------------------------------------|
| Mild | 1 or 2 Organs involved with no more than score 1 plus |
| | Lung score 0. |
| Moderate | 3 or More organs involved with no more than score 1 OR |
| | At least 1 organ (not lung) with a score of 2 OR |
| | Lung score 1 |
| Severe | At least 1 organ with a score of 3 |
| | OR |
| | Lung score of 2 or 3 |

**Notes**: GVHD=graft-versus-host disease; In skin: higher of the 2 scores to be used for calculating global severity. In lung: FEV1 is used instead of clinical score for calculating global severity. If the entire abnormality in an organ is noted to be unequivocally explained by a non-GVHD documented cause, that organ is not included for calculation of the global severity. If the abnormality in an organ is attributed to multifactorial causes (GVHD plus other causes) the scored organ will be used for calculation of the global severity regardless of the contributing causes (no downgrading of organ severity score). \* Jagasia MH, Greinix HT, Arora M, et al. National Institutes of Health Consensus Development Project on Criteria for Clinical Trials in Chronic Graft-versus-Host Disease: I. The 2014 Diagnosis and Staging Working Group report. Biol Blood Marrow Transplant. 2015;21(3):389-401.

## Appendix 5. The table of study procedure

| | 6-month follow-up | | | | | × | | × | | × | × |
|---|---|---|---|---|---|---|---|---|---|---|---|
| | 6-month | | | | | ^ | | ^ | | ^ | ^ |
| | 28 | | | | × | × | × | × | | × | × |
| | 27 | | | | | × | | | | × | × |
| | 56 | | | | | × | | | | × | × |
| | 25 | | | | | × | × | | | × | × |
| | 24 | | | | | × | | | | × | × |
| | 23 | | | | | × | | | | × | × |
| | 22 | | | | | × | × | | | × | × |
| | 21 | | | | | × | | | | × | × |
| | 20 | | | | | × | | | | × | × |
| | 19 | | | | | × | × | | | × | × |
| | 18 | | | | | × | | | | × | × |
| eriod | 17 | | | | | × | | | | × | × |
| Study Period | 16 | | | | | × | × | | | × | × |
| ν | 15 | | | | | × | | | | × | × |
| | 14 | | | | | × | | | | × | × |
| | 13 | | | | | × | × | | | × | × |
| | 12 | | | | | × | | | | × | × |
| | 11 | | | | | × | | | | × | × |
| | 10 | | | | | × | × | | | × | × |
| | 6 | | | | | × | | | | × | × |
| | ∞ | | | | | × | | | | × | × |
| | 7 | | | | | × | × | | | × | × |
| | 9 | | | | | × | | | | × | × |
| | 2 | | | | | × | | | | × | × |
| | 4 | | | | | × | × | | | × | × |
| | m | | | | | × | | | × | | × |
| | 2 | | | | | × | | | × | | × |
| | 1 | | | | | × | × | | × | | × |
| Screening | -3 — -1 | × | × | × | × | × | × | × | | | |
| Procedure | Day | Patient<br>Consent<br>Form | Demographic<br>data | General<br>information | Physical examination | Peripheral<br>blood counts | renal and<br>liver function<br>test | Bone marrow examination | Decitabine | rhTPO | Conventional<br>therapy |
| Proc | | | | | | | oterode<br>itenime | | ţи | tme | Trea |

#### Appendix 6: Patient consent form for study participation

| Title: Low-dose decitabine for refractory prolonged isolated | | |
|---|---|---|
| thrombocytopenia af | thrombocytopenia after hematopoietic cell transplantation | |
| Investigator OR | Study Sit | е |
| institution Name | | |
| Patient Name | | |
| Please <b>tick</b> each box | Please <b>tick</b> each box below □ if you have known the corresponding | |
| statement. | | |
| (to be completed by the patient) | | |

#### ☐ What you should know about a research study

Someone will explain this research study to you.

- A research study is something you volunteer for.
- Presence or absence of participation in the research study is up to you.
- You can choose not to take part in the research study.
- You can agree to take part now and later change your mind.
- Whatever you decide it will not be held against you.
- You can feel free to ask all the questions that you want before you decide.

#### ☐ What is the purpose of this study?

Refractory prolonged isolated thrombocytopenia (RPIT), a frequent complication after hematopoietic stem cell transplantation (HCT), is associated with significantly adverse outcomes. It is urgent to explore effective agents that can promote the platelet recovery and prevent potentially fatal bleeding complications. We previously reported a pilot study which described the effectiveness of low-dose decitabine for increasing platelet counts in transplant recipients with RPIT by increasing the number of marrow megakaryocyte.

To further validate the efficacy and safety of low-dose decitabine for RPIT and to preliminarily explore the potential mechanisms, this prospective, open-label, three-arm, randomized clinical trial is conducted.

#### ☐ Why have I been chosen?

We are inviting patients who

Platelet count < 30 × 10<sup>9</sup>/L for more than 60 days post-HCT;

- Recovered neutrophil and hemoglobin concentrations;
- Donor chimerism >95% detected by short-tandem repeat-polymerase chain reaction;
- No response to conventional treatments for thrombocytopenia (rhTPO, immunoglobulin, rituximab and glucocorticoid, either alone or in combination) for a duration of at least 4 weeks.

#### ☐ Do I have to take part?

- Participation in the study is entirely voluntary.
- You will be given sufficient time to consider whether you want to participate in the study.
- Non-participation in the study will not affect your future care that you will receive from your medical and nursing team in our hospital.
- If you decide to join the study, you will be asked to sign an informed consent form.
- You are free to withdraw from this research at any time and without giving a reason. Any of your current medical care and future treatment in our hospital will not be affected.

#### ☐ What will happen to me if I take part?

All patients who agree to take part and provide a written informed consent form will be included into this study.

If you are included in this research, you will be randomly assigned into the one of three treatment group. Randomization means that neither you nor your doctor will be able to select which treatment you will receive. We will use a computer to allocate you to one of this three groups with equal chances of each treatment approach being the one you will receive. This procedure will ensure that the number of patients in each of the three treatment groups is similar.

➤ If you are assigned in the group A:

You will be treated with decitabine (15 mg/m² daily intravenously for consecutive 3 days (day 1 - day 3)) plus recombinant human thrombopoietin (300 U/kg.d from day 4 to day 28);

➤ If you are assigned in the group B:

You will be treated with decitabine alone (15 mg/m<sup>2</sup> daily intravenously for consecutive 3 days);

If you are assigned in the group C:

You will be treated with conventional treatments as usual.

Your doctors will introduce the detailed treatment procedures to you. You are free to ask any question about the treatments you may have.

#### ☐ How long will I be in the study

If you participate in this study, you will receive <u>1</u> therapy for 4 weeks. Follow up will continue indefinitely, for as long as <u>6</u> months or longer.

You can stop participating at any time. However, if you decide to stop participating in the study, we encourage you to talk to the researcher and your regular doctor first.

#### ☐ What are the risks of the study?

#### Potential adverse event of decitabine includes:

#### • Myelosuppression:

Neutropenia related infections, fever;

Bleeding: ecchymosis, petechial, haematemesis, hemoptysis, melena, hematuresis, etc;

Weary, somnolence, pale, etc (due to anemia);

#### Other non-hematological toxicity:

Liver dysfunction;

Renal dysfunction;

#### Drug allergy

Erythra, edema, pruritus, swelling, etc

#### Potential adverse event of rhTPO includes:

Thrombosis, injection site reaction (subcutaneous scleroma, fat atrophy, ache, etc), drug allergy.

#### Others:

There also may be other unexpected complications or discomforts that we cannot predict.

Your doctors will do their best to prevent complications and to treat them if occur. You will receive the best medical care available during and after the study and in the unlikely event of an injury arising from taking part in this study, you will be provided with the necessary care.

#### □Are there benefits you to taking part in the study?

You'll get free treatment of rhTPO (Group A) and free test of blood and bone marrow (all participants). Another possible benefit you may experience from this

research includes recovery of your platelet level and prolongation of survival time. However, there is no guarantee that each patient will benefit from the treatment in this research.

Furthermore, the results obtained from this study may be useful in guiding the treatment for patients with such disease in the future.

#### ☐ What are my responsibilities in this study?

If you choose to take part in this study, you will need to:

- Keep your study appointments.
- Tell your doctor about:
- · All medications and supplements you are taking;
- Any discomforts or complications you suspect;
- Any doctors' visits or hospital stays outside of this study;
- Whether you have been or are currently in another research study.

#### ☐ How will my privacy be protected?

Your health information, such as your response to cancer treatment, results of study tests, and medicines you took, will be kept by the data center of this research. This information is strictly confidential. However, your name and contact information will not be put in the database. If information from this study is published or presented at scientific meetings, there will be no personally identifiable information.

#### ☐ What happens if I change my mind during the study?

We would certainly recommend that you continue the study, however, participation in the study is voluntary and you may stop the participation at any time that you wish without losing any of your rights as a patient here. Your treatment at our hospital will not be affected in any way. The PI of this study also has the right to withdraw patients from the study if he feels that the withdrawal is in your best interests. Your follow-up information will still be kept by doctor after you have stopped participating in the research.

#### ☐ Who is organizing the research?

The study is organized by the The First Affiliated Hospital of Soochow University, Suzhou 215006, China. There are five other participating institutes including Nanfang Hospital, Southern Medical University, Guangzhou 510515, China, Fujian Institute of Hematology, Fuzhou 350001, China, Children's Hospital of Soochow University, Suzhou 215025, China, Hebei Yanda Lu

| Daopei Hospital, Langfang 065201, China and Rui Jin Hospital, Shanghai Jiao<br>Tong University School of Medicine, Shanghai 200025, China. | |
|---|---|
| □Whom do I call if I have questions or pr | oblems? |
| For information about your disease and resecontact: | earch-related injury, you may |
| Name (institution) : | Telephone Number: |
| For information about this study, you may co | ontact: |
| Name (institution) : Telephone Number: | |
| For information about your rights as a resea | rch subject, you may contact: |
| Name (institution) : | Telephone Number: |

#### Signature page

I have read all the above, asked questions, and received answers concerning areas I did not understand. I have had the opportunity to take this consent form home for review or discussion.

I willingly give my consent to participate in this program. Upon signing this form I will receive a copy. I may also request a copy of the protocol (full study plan).

| Patient | Name | Date |
|-----------|---------|--------|
| signature | (print) | signed |

## Investigator (institution) Statement and Signature to be completed by the person taking consent

I have discussed this clinical research study with the patient and/or his or her authorized representative using a language that is understandable and appropriate. I believe that I have fully informed the participant of the nature of this study and the possible benefits and risks of taking part. I believe the participant has understood this explanation.

| Investigator OR | Name | Date |
|-----------------------|---------|--------|
| institution signature | (print) | signed |